CLINICAL TRIAL: NCT06642688
Title: Comparison Of Spinal Manipulation Applied to the Cervical Spine and Sacroiliac Joints With Pedobarographic Analysis and It's Immediate Effect on the Autonomic Nervous System in Healthy Individuals
Brief Title: Immediate Effect of Cervical and Sacroiliac Manipulation on the Autonomic Nervous System and Balance
Acronym: CSMPAANS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SEFA HAKTAN HATIK (Other)
Responsible Party: Sponsor-Investigator, SEFA HAKTAN HATIK, Asst. Professor, Sinop University
Organization: Sinop University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: CMT0006
Record Dates: First submitted 2024-10-09; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Neuromuscular Subluxation of Joint; Manual Therapy; Autonomic Nervous System Activity
Keywords: Chiropractic; Cervical Spine; Sacroiliac Joint; Autonomic Nervous System; Pedobarographic Analysis

STUDY DESIGN:
Intervention Model Description: Ninety-six participants who met the inclusion criteria were enrolled in the study and were divided into three groups: the sacroiliac joint manipulation group (n=32), the cervical manipulation group (n=32), and the control group (n=32). Sacroiliac joint manipulation was performed in the lateral decubitus position, while cervical manipulation was applied in the supine position, and no treatment was administered to the control group. All measurements were repeated before and immediately after the manipulations. The Mann-Whitney U test was used to determine whether the scores differed according to a dichotomous variable, while the Kruskal-Wallis test was used for variables with more than two categories. In cases where significant differences were found between categories, the Mann-Whitney U test with multiple comparisons was used to identify the source of the difference between the pairwise groups.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Sacroiliac Joint Manipulation Group (Experimental): Sacroiliac joint manipulation was performed on this group in the lateral decubitus position.
  Interventions: Other: Sacroiliac Joint Manipulation
- Cervical Joint Manipulation Group (Experimental): Cervical joint manipulation was performed on this group in the supine position.
  Interventions: Other: Cervical Spine Manipulation
- Control Group (No Intervention): This group did not undergo any interventions.

INTERVENTIONS:
Other: Sacroiliac Joint Manipulation — The patient was asked to tie his arms while he was in the side lying position. The patient's upper knee was flexed and positioned such that it was placed in the popliteal fossa of the lower knee, while the lower knee was in full extension. Pushing maneuver was performed with HVLA from posterior to anterior and from medial to lateral with pelvic rotation. The contact point of the sacroiliac joint was PSIS.
  Arms: Sacroiliac Joint Manipulation Group
Other: Cervical Spine Manipulation — Cervical SM was applied supine to restrictions found on motion palpation, according to the technique described by Bergmann and Peterson28 The participant's head and neck were simultaneously rotated and laterally flexed over the contact point-specifically, the posterior supramastoid groove or zygomatic arch (C0-C1), the posterior aspect of the transverse process (C1-C2), or the posterior articular pillar of superior vertebrae (C2-C7) -to the end of passive ROM. Thereafter, a high-velocity, low-amplitude thrust was delivered in the direction of restricted movement. Participants with more ROM restriction in the lateral plane were given more lateral-to-medial directed thrusts; participants with more restriction in rotation were given thrusts in the direction of restricted axial rotation; and participants with more restriction in extension were given more anteriorly directed thrusts.
  Arms: Cervical Joint Manipulation Group

SUMMARY:
The aim of this study is to investigate the immediate effects of high-velocity low-amplitude (HVLA) chiropractic manipulation on the autonomic nervous system and baropodometric parameters. The effects of different manipulation techniques on pedobarographic analysis and the autonomic nervous system were examined.

DETAILED DESCRIPTION:
Ninety-six individuals who met the inclusion criteria participated in the study. The participants were divided into three groups: the sacroiliac joint manipulation group (n=32), the cervical manipulation group (n=32), and the control group (n=30). No treatment was administered to the control group, while sacroiliac joint manipulation and cervical manipulation were applied to the sacroiliac joint manipulation group and the cervical manipulation group, respectively. Autonomic nervous system activity was assessed using the Polar H-10 device, pedobarographic analysis was performed using the METISENS pedobarographic evaluation device, and blood pressure and pulse were measured manually from the left arm using a sphygmomanometer. A 30-minute waiting period was used during the evaluation of the control group. A significance level of p<0.05 was considered

ELIGIBILITY:
Inclusion Criteria:

* Willingness to participate voluntarily.
* Signed informed consent form.
* Age between 18 and 35 years.
* No contraindications for chiropractic practices.

Exclusion Criteria:

* History of orthopedic disabilities related to the lower extremity.
* Ankylosing spondylitis, rheumatoid arthritis.
* History of foot sprain/strain within the past six months.
* Presence of pathologies in the lumbar and sacroiliac regions (herniated discs, spondylosis, spondylolisthesis).
* History of cardiovascular and respiratory diseases.
* Psychiatric disorders such as psychosis and depression.
* Radicular root compressions causing progressive neurological deficits.
* Bleeding/coagulation disorders and receiving anticoagulant treatment.
* Acute fractures and orthopedic trauma.
* Spinal cord tumors and meningeal tumors.
* Intraosseous infections and acute inflammation, such as osteomyelitis.
* Cauda equina syndrome.
* Intracanicular hematomas.
* Spinal cord hematomas in the spine.
* Basilar invagination of the upper cervical region.
* Aneurysmal bone cysts, osteoid osteomas, osteolastomas, giant cell bone tumors.
* Post-surgical fixation prostheses.
* Neoplastic diseases in muscles or other tissues.
* Lhermitte's sign.
* Syringomyelia.
* Vertebral dislocations or hypermobile joints.
* Advanced osteoporosis.
* Vertebrobasilar insufficiency.

Criteria for Withdrawal from the Study:

* Pregnancy or suspicion of pregnancy.
* The volunteer's desire to discontinue participation in the study.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 96 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Evaluation of Autonomic Nervous System | In the manipulation groups, measurements were repeated immediately after the manipulation, while in the control group, the initial measurements were repeated 30 minutes later.
  The assessment of the autonomic nervous system was conducted using the Polar H10 device, which is a high-accuracy, gold-standard HRV sensor that comes with a chest-worn strap. The device can connect to multiple components via Bluetooth and ANT+. This device facilitates the measurement of heart rate variability (HRV), R-R intervals, RMSSD (an instantaneous assessment of the parasympathetic system), LF Power (activation of the sympathetic nervous system), HF Power (activation of the parasympathetic nervous system), HF band, and LF/HF ratio (sympathetic-vagal balance).
  For data analysis, the Elite HRV software supported by the device is utilized. Measurements are conducted while the participant is seated and last approximately one minute. To ensure accurate measurements, it is necessary to moisten the electrode surface before each measurement. During the assessment, the participant should not speak or move
Evaluation of Blood Pressure | In the manipulation groups, measurements were repeated immediately after the manipulation, while in the control group, the initial measurements were repeated 30 minutes later.
  Blood pressure of the participants were evaluated with a manual sphygmomanometer on the left arm.
Analysis of Pedobarographic Data | In the manipulation groups, measurements were repeated immediately after the manipulation, while in the control group, the initial measurements were repeated 30 minutes later.
  The analysis of pedobarographic data was conducted using METISENS pedobarographic assessment devices. During the measurements of pressure analysis in individuals participating in our study, static conditions were maintained, and the load distribution on both the right and left feet, as well as the loads on the anterior and posterior aspects of the foot (%), were reported. Pressure analyses were determined using the Metisens Baropodometric Analysis software, which is the proprietary software that operates in conjunction with the Metisens Pedobarographic Assessment Device (It is not possible to separate these measurements as the device takes all measurements and provides a total analysis.)
Evaluation of Pulse | In the manipulation groups, measurements were repeated immediately after the manipulation, while in the control group, the initial measurements were repeated 30 minutes later.
  The pulse of the participants were evaluated with a manual sphygmomanometer on the left arm.

CONTACTS AND LOCATIONS:
Overall Officials: SEFA H HATIK, Asst. Prof., Principal Investigator — Sinop University
Locations (1):
- Sinop University, Sinop, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No